CLINICAL TRIAL: NCT01210144
Title: Open Label Pilot Study on Gene Expression Profiling of the Endometrial Tissue in Patients Undergoing Assisted Reproductive Technology [ART: In Vitro Fertilization (IVF)/ Intracytoplasmic Sperm Injection (ICSI)] With GONAL-f®
Brief Title: EXpression PRofile Endometrium Samples Study
Acronym: EXPRESS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated due to recruitment failure
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono S.A.S, France (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMP 28364; 2007-003938-41 (EudraCT Number)
Record Dates: First submitted 2010-08-11; First posted 2010-09-28 (Estimated); Results first posted 2012-11-14 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: In Vitro Fertilization
Keywords: Infertility; Gonal-f; gene expression; Assisted Reproductive Technologies; Follitropin alfa; endometrium
MeSH Terms: conditions — Infertility | interventions — Glycoprotein Hormones, alpha Subunit; follitropin alfa; Chorionic Gonadotropin; Ovidrel; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gonal-f® + Ovitrelle® + Long Agonist Protocol (Experimental)
  Interventions: Drug: Gonal -f® [r-hFSH]; Drug: Ovitrelle® [r-hCG alfa]; Drug: Gonadotropin-releasing hormone (GnRH) Agonist
- Gonal-f® + Ovitrelle® + Multi-dose Antagonist Protocol (Experimental)
  Interventions: Drug: Gonal -f® [r-hFSH]; Drug: Ovitrelle® [r-hCG alfa]; Drug: Gonadotropin-releasing hormone (GnRH) Antagonist

INTERVENTIONS:
Drug: Gonal -f® [r-hFSH] — On Day 2 of the menstrual cycle, a pre-defined fixed dose of 150 International Units (IU) per day of recombinant human follicle stimulating hormone (r-hFSH) will be administered until follicles are recruited and developed.
  Other Names: Gonal-f®; Follitropin Alfa
Drug: Ovitrelle® [r-hCG alfa] — Ovulation triggering will be performed using a single injection of 250 microgram (mcg) recombinant human chorionic gonadotropin (r-hCG) alfa as soon as follicles satisfy the criteria for follicular development, that is at least 3 follicles greater than (>) 16 millimeter (mm), and with estradiol (E2) > 1 microgram per liter (mcg/L) if gonadotropin releasing hormone (GnRH) agonist will be used.
  Other Names: Ovitrelle®; Ovidrel®
Drug: Gonadotropin-releasing hormone (GnRH) Agonist — To prevent premature ovulation in participants undergoing a controlled ovarian stimulation (COS), 0.1 milligram (mg) GnRH agonist daily will be given after endometrial biopsy, 7 days after the peak day of luteinizing hormone (Day LH + 7) as per summary of product characteristics (SmPC), in long agonist protocol.
  Arms: Gonal-f® + Ovitrelle® + Long Agonist Protocol
Drug: Gonadotropin-releasing hormone (GnRH) Antagonist — To prevent premature ovulation in participants undergoing a COS, 0.25 mg GnRH antagonist daily will be given from Day 6 of Gonal-f® stimulation treatment as per SmPC, in multi-dose antagonist protocol.
  Arms: Gonal-f® + Ovitrelle® + Multi-dose Antagonist Protocol

SUMMARY:
This is a Phase IV, pilot, open-label, national, multi-centric study planned to determine the gene expression profiles and histologic changes of the endometrial tissue before and after stimulation with Gonal-f®. Physicians are interested in identifying predictive genetic markers in assisted reproductive technologies (ART) in addition to the clinical predictive factors already known. Among those predictive factors, the state of the endometrium is considered as an important implantation determining factor for which pharmacogenomic research is of great interest.

The direct benefits of this study will be to know whether the endometrial gene expression profile is modified in response to stimulation treatment and have an impact or not on the endometrial tissue receptivity. The potential benefits of this study could be to assess the therapy optimization based on individual treatment response and gene expression profile compared to group treatment response in infertile women and prediction of response to therapy based on gene expression profiling before and after Gonal-f® stimulation in infertile women.

DETAILED DESCRIPTION:
This is a pilot open-label, national, multi-centre, Phase IV trial. This trial will be conducted with outpatients. Once subject has met all eligibility criteria, she will be treated with Gonal-f® prefilled pen and will receive on a randomization basis the GnRH agonist or antagonist. The follicle stimulating hormone (FSH) stimulation will start on day 2 of the menstrual cycle with a pre-defined fixed dose of 150 IU per day until follicles are recruited and developed. Dose adjustment will be allowed strictly in case of risk of ovarian hyperstimulation syndrome (OHSS). Ovulation triggering will be performed using a single injection of 250 mcg Ovitrelle®.

Ultrasound scans (US) will be performed concomitantly with hormonal assessment at each visit. Ovulation will be triggered as soon as there are at least 3 follicles > 16 mm, and with E2 > 1 mcg/L if agonist used. Oocyte retrieval, in vitro fertilization (IVF) or intra-cytoplasmic sperm injection (ICSI) and blastocyst transfer will be performed as per centre's standard practice. Vaginal progesterone will be administered in the luteal phase for all subjects (600 milligram per day [mg/d]).

Hormonal assessment and endometrial biopsy will be performed on:

* Day Luteinizing Hormone+7 ("LH+7") of the previous spontaneous cycle
* Day of Oocyte Retrieval (OR) of the stimulated cycle
* Day "OR+5 or 6" (biopsy performed only in subjects that did not have blastocyst(s) transfer).

Gene expression profiling will be carried out on ribonucleic acid (RNA) from endometrial tissue. As the main objective of this trial is to determine the gene expression profiles of endometrial tissue before and after controlled ovarian stimulation with Gonal-f®, a minimum of 2 endometrial samples per subject will be collected, 1 at day LH+7 of spontaneous cycle and 1 after the stimulation, on the day of OR.

The subjects will be followed up until 15 days after the last injection of Investigational Medicinal Products (IMPs) for the safety assessment. For subjects who will have blastocyst implantation, the pregnancy outcomes will be recorded until 12 weeks of gestation if a pregnancy is ongoing up to that period.

OBJECTIVES

Primary objective:

* To determine the gene expression profile and histological changes of endometrial tissue before (at day LH + 7 of spontaneous cycle) and after stimulation with Gonal-f® (Day of OR: 36 +/- 2 hours post r-hCG administration) in Assisted Reproductive Technology (ART) [IVF/ICSI]

Secondary objectives:

* To correlate the gene expression profile of the endometrial tissue at Day LH + 7 of the spontaneous cycle with the blastocyst implantation rate in subjects undergoing ART with Gonal-f®
* To correlate the gene expression profile and histological changes in endometrial tissue before and after stimulation by Gonal-f® with the "down regulation" protocol used (agonist or antagonist) and fertilization mode, IVF/ICSI
* To correlate the gene expression profile and histological changes in endometrial tissue before and after stimulation by Gonal-f® according to the hormonal status of subjects
* To characterize the gene expression profile and histology of endometrial tissue after stimulation with Gonal-f in subjects without blastocyst during the theoretical window of implantation (OR + 5 or 6 days)
* To characterize the gene expression profile and histology of endometrial tissue of good and poor responders to stimulation with Gonal-f® on the Day of OR (response being based on the following criteria):

  1. Quantity of mature oocytes retrieved:

     * Poor responders: 5 mature oocytes or less
     * Good responders: more than 8 mature oocytes
  2. Quantity of Gonal-f® used

ELIGIBILITY:
Inclusion Criteria:

* Infertile female or infertile male. Infertile female means diverse infertility etiologies including tubal disease (excepting hydrosalpinx) and so called "unexplained infertility"
* Suitable for ART: IVF undergoing first or second attempt, ICSI undergoing first attempt
* 18-35 years old, body mass index (BMI) less than or equal to 27 kilogram per square meter (kg/m^2), non smoking
* Normal ovarian status (FSH less than or equal to 9.45 International Units per Liter [IU/L], E2 less than or equal to 40 picogram per milliliter [pg/mL], Anti-Mullerian Hormone [AMH] greater than or equal to 18 picomole/liter [pmol/L]; within normal laboratory range values, normal ovaries sonography and uterine echo doppler)
* No history of active genito-urinary infection
* Normal thyroid function (or adequate substitution for at least 3 months)
* Negative cervical papanicolaou test within the last 12 months prior to study entry
* No hormonal therapy, including gonadotropins and progesterone, for at least 2 months prior to the study
* In couple with female infertility, male partner with normal sperm or moderate oligoasthenospermia in semen analysis and negative semen culture less than 6 months at the study entry
* Willingness and ability to comply with the protocol for the duration of the study
* Written informed consent prior to any study related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to their future medical care

Exclusion Criteria:

* Subjects with ongoing pregnancy, any pregnancy within 3 months prior to study entry, or any contraindication to pregnancy or carrying pregnancy to term
* Subjects with uterine malformation, diethylstilbestrol syndrome, adenomyosis, synechia
* Subjects with history of previous OHSS
* Subjects with polycystic ovarian syndrome (PCOS) according to the revised Rotterdam Consensus 2003
* Subjects with extra-uterine pregnancy during the previous 3 months
* Subjects with recurrent miscarriages (early or late, more than 2)
* Subjects having known infection with human immunodeficiency virus (HIV), hepatitis B or C virus, for subject or partner
* Subjects with abnormal gynecological bleeding of undetermined origin
* Subjects with history of major thromboembolic disease
* Subjects with endometriosis
* Subjects with presence or history of malignant tumors and related treatment
* Subjects with clinically significant systemic disease or clinically significant abnormal hematology, chemistry, or urinalysis results at screening
* Subjects with known allergy or hypersensitivity to Gonal-f® or Ovitrelle®
* Subjects with any active substance abuse or history of drug, medication or alcohol abuse in the past 5 years
* Subjects who have participated within 3 months prior to study entry in another clinical trial

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2008-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Paris, France

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 27 participants were enrolled in the study, out of which 2 participants withdrew the consent and 1 participant was excluded since endometrial biopsy was not possible.
Groups:
- Gonal-f® + Ovitrelle® (Long Agonist Protocol): Participants received 150 International Units (IU) per day of recombinant human follicle stimulating hormone (r-hFSH, Gonal-f®) subcutaneously (sc) starting from Day 2 of menstrual cycle until follicles were recruited and developed. Ovulation triggering was performed with a single dose of 250 microgram (mcg) recombinant human chorionic gonadotropin alfa (r-hCG alfa, Ovitrelle®) sc, as soon as follicles satisfied the criteria for follicular development (at least 3 follicles greater than [>] 16 millimeter [mm], and with estradiol [E2] >1 microgram per liter [mcg/L]). To prevent premature ovulation in participants undergoing a controlled ovarian stimulation (COS), 0.1 milligram (mg) gonadotropin-releasing hormone (GnRH) agonist daily was started after endometrial biopsy, 7 days after the peak day of luteinizing hormone (Day LH + 7) as per summary of product characteristics (SmPC), in long agonist protocol.
- Gonal-f® + Ovitrelle® (Multi-dose Antagonist Protocol): Participants received 150 IU per day of r-hFSH (Gonal-f®) sc starting from Day 2 of menstrual cycle until follicles were recruited and developed. Ovulation triggering was performed with a single dose of 250 mcg r-hCG alfa (Ovitrelle®) sc, as soon as follicles satisfied the criteria for follicular development (at least 3 follicles >16 mm). To prevent premature ovulation in participants undergoing a COS, 0.25 mg GnRH antagonist daily was started from Day 6 of Gonal-f® stimulation treatment as per SmPC, in multi-dose antagonist protocol.
Period: Overall Study
Arm/Group | Gonal-f® + Ovitrelle® (Long Agonist Protocol) | Gonal-f® + Ovitrelle® (Multi-dose Antagonist Protocol)
Started | 13 | 11
Completed | 10 | 11
Not Completed | 3 | 0
Not completed — Lack of ovarian response | 1 | 0
Not completed — No fertilization | 1 | 0
Not completed — No transfer | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Gonal-f® + Ovitrelle® (Long Agonist Protocol): Participants received 150 International Units (IU) per day of recombinant human follicle stimulating hormone (r-hFSH, Gonal-f®) subcutaneously (sc) starting from Day 2 of menstrual cycle until follicles were recruited and developed. Ovulation triggering was performed with a single dose of 250 microgram (mcg) recombinant human chorionic gonadotropin alfa (r-hCG alfa, Ovitrelle®) sc, as soon as follicles satisfied the criteria for follicular development (at least 3 follicles greater than [>] 16 millimeter [mm], and with estradiol [E2] >1 microgram per liter [mcg/L]). To prevent premature ovulation in participants undergoing a controlled ovarian stimulation (COS), 0.1 milligram (mg) GnRH agonist daily was started after endometrial biopsy, 7 days after the peak day of luteinizing hormone (Day LH + 7) as per summary of product characteristics (SmPC), in long agonist protocol.
- Total: Total of all reporting groups
Arm/Group | Gonal-f® + Ovitrelle® (Long Agonist Protocol) | Gonal-f® + Ovitrelle® (Multi-dose Antagonist Protocol) | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (4.2) | 31.0 (4.4) | 30.4 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Gene Expression of the Endometrium Following 1 Cycle With Gonal-f®
Description: A list of genes based on gene expression profiling carried out on ribonucleic acid (RNA) extracted from endometrial tissue. The expression of messenger ribonucleic acid (mRNA) in endometrial tissue was measured by using microarrays such as the Affymetrix® GeneChip HG-U133 plus 2.0 array or equivalent.
Time Frame: Day of Oocyte Retrieval (36 +/- 2 hours post r-hCG administration) after COS by Gonal-f®
Population: Data were not analyzed for both agonist and antagonist protocol as total, which was the primary objective, since gene expression of the endometrium could not be performed due to poor quality of biopsy samples and poor recruitment in the study.
Groups:
- Gonal-f® + Ovitrelle®: Participants received 150 IU per day of r-hFSH (Gonal-F®) sc starting from Day 2 of menstrual cycle until follicles were recruited and developed. Ovulation triggering was performed with a single dose of 250 mcg r-hCG alfa (Ovitrelle®) sc, as soon as follicles satisfied the criteria for follicular development (at least 3 follicles >16 mm [for both long agonist and multi-dose antagonist protocol], and with E2>1 mcg/L [for long agonist protocol]). To prevent premature ovulation in participants undergoing a controlled ovarian stimulation, either 0.1 mg GnRH agonist daily was started after endometrial biopsy, 7 days after the peak day of luteinizing hormone (Day LH + 7) in long agonist protocol or 0.25 mg GnRH antagonist daily was started from Day 6 of GONAL-f® stimulation treatment in multi-dose antagonist protocol, as per SmPC.
Arm/Group | Gonal-f® + Ovitrelle®
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants With a Specific Histological Pattern of the Endometrium Following 1 Cycle With Gonal-f®
Description: Participants with each histological pattern of endometrium were analyzed. Histological patterns included: Proliferative phase (described as the endometrial on the first two weeks after the menstruation [or before ovulation]), Early secretory phase (first step of the secretory phase, located at the Day 16-18 of the cycle) and Intermediate secretory phase (secretory phase located at the Day 20-22 of the cycle and describes endometrial closer to the implantation phase).
Time Frame: Day of Oocyte Retrieval (36 +/- 2 hours post r-hCG administration) after COS by Gonal-f®
Population: Intention-to-Treat (ITT) population: participants who received at least 1 dose of study drug. "N" (number of participants analyzed) signifies participants evaluable for this measure. Results for both agonist and antagonist protocol are presented as total since assessment of histological pattern for whole study population was the primary objective.
Measure: Number; unit: participants
Arm/Group | Gonal-f® + Ovitrelle®
Number analyzed (Participants) | 23
participants
  Proliferative phase | 2
  Early secretory phase | 15
  Intermediate secretory phase | 6

3. Secondary Outcome: Gene Expression of the Endometrium in Participants With or Without Blastocyst Transfer
Description: A list of genes based on gene expression profiling carried out on RNA extracted from endometrial tissue. The expression of mRNA in endometrial tissue was measured by using microarrays such as the Affymetrix® GeneChip HG-U133 plus 2.0 array or equivalent.
Time Frame: Day of Oocyte Retrieval (36 +/- 2 hours post r-hCG administration) after COS by Gonal-f®
Population: Data were not analyzed because gene expression of the endometrium could not be performed due to poor quality of biopsy samples and poor recruitment in the study.
Arm/Group | Gonal-f® + Ovitrelle® (Long Agonist Protocol) | Gonal-f® + Ovitrelle® (Multi-dose Antagonist Protocol)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Gene Expression of the Endometrium Following 1 Cycle With Gonal-f® in Participants Having Undergone Agonist or Antagonist Protocol
Description: as for outcome 3
Time Frame: Day of Oocyte Retrieval (36 +/- 2 hours post r-hCG administration) after COS by Gonal-f®
Population: as for outcome 3
Arm/Group | Gonal-f® + Ovitrelle® (Long Agonist Protocol) | Gonal-f® + Ovitrelle® (Multi-dose Antagonist Protocol)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With a Specific Histological Pattern of the Endometrium Following 1 Cycle With Gonal-f® and Having Undergone Agonist or Antagonist Protocol
Description: Participants with each histological pattern of endometrium were analyzed. Histological patterns included: Proliferative phase (described as the endometrial on the first two weeks after the menstruation [or before ovulation]), Early secretory phase (first step of the secretory phase, located at the Day 16-18 of the cycle), Intermediate secretory phase (secretory phase located at the Day 20-22 of the cycle and describes endometrial closer to the implantation phase).
Time Frame: Day of Oocyte Retrieval (36 +/- 2 hours post r-hCG administration) after COS by Gonal-f®
Population: ITT population included those participants who received at least one dose of study medication. Here "N" (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Gonal-f® + Ovitrelle® (Long Agonist Protocol) | Gonal-f® + Ovitrelle® (Multi-dose Antagonist Protocol)
Number analyzed (Participants) | 12 | 11
participants
  Proliferative phase | 1 | 1
  Early secretory phase | 8 | 7
  Intermediate secretory phase | 3 | 3

6. Secondary Outcome: Gene Expression in Participants Without Blastocyst Transfer
Description: as for outcome 3
Time Frame: Day 5 or 6 (window of implantation) after Oocyte Retrieval
Population: as for outcome 3
Arm/Group | Gonal-f® + Ovitrelle® (Long Agonist Protocol) | Gonal-f® + Ovitrelle® (Multi-dose Antagonist Protocol)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With a Specific Histological Pattern of the Endometrium in Participants Without Blastocyst Transfer
Description: as for outcome 5
Time Frame: Day 5 or 6 (window of implantation) after Oocyte Retrieval
Population: ITT population: participants who received at least one dose of study medication. "N" (number of participants analyzed) signifies participants who were evaluable for this measure. Data were not analyzed for Gonal-f® + Ovitrelle® (Multi-dose Antagonist Protocol) group because there were no participants without blastocyst transfer in this group.
Measure: Number; unit: participants
Arm/Group | Gonal-f® + Ovitrelle® (Long Agonist Protocol) | Gonal-f® + Ovitrelle® (Multi-dose Antagonist Protocol)
Number analyzed (Participants) | 2 | 0
participants
  Proliferative phase | 0 |
  Early secretory phase | 0 |
  Intermediate secretory phase | 2 |

8. Secondary Outcome: Gene Expression in Participants With Good or Poor Response to Gonal-f®
Description: A list of genes based on gene expression profiling carried out on RNA extracted from endometrial tissue. The expression of mRNA in endometrial tissue was measured by using microarrays such as the Affymetrix® GeneChip HG-U133 plus 2.0 array or equivalent. Participants with poor response: 5 mature oocytes or less; participants with good response: more than 8 mature oocytes.
Time Frame: Day of Oocyte Retrieval (36 +/- 2 hours post r-hCG administration) after COS by Gonal-f®
Population: as for outcome 3
Arm/Group | Gonal-f® + Ovitrelle® (Long Agonist Protocol) | Gonal-f® + Ovitrelle® (Multi-dose Antagonist Protocol)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants With a Specific Histological Pattern of the Endometrium in Participants With Good or Poor Response to Gonal-f®
Description: Participants with each histological pattern of endometrium were analyzed. Histological patterns included: Proliferative phase (described as the endometrial on the first two weeks after the menstruation [or before ovulation]), Early secretory phase (first step of the secretory phase, located at the Day 16-18 of the cycle), Intermediate secretory phase (secretory phase located at the Day 20-22 of the cycle and describes endometrial closer to the implantation phase). Participants with poor response: 5 mature oocytes or less; participants with good response: more than 8 mature oocytes.
Time Frame: Day of Oocyte Retrieval (36 +/- 2 hours post r-hCG administration) after COS by Gonal-f®
Population: Data for histological pattern of the endometrium in participants with good or poor response to Gonal-f were not summarized because the number of participants in each group with respect to ovarian response were too low.
Arm/Group | Gonal-f® + Ovitrelle® (Long Agonist Protocol) | Gonal-f® + Ovitrelle® (Multi-dose Antagonist Protocol)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 15 days after the last Investigational Medicinal Product (IMP) administration or early termination
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerge or worsen relative to baseline during a clinical study with an IMP, regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Gonal-f® + Ovitrelle® (Long Agonist Protocol) | Gonal-f® + Ovitrelle® (Multi-dose Antagonist Protocol)
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 2/13 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gonal-f® + Ovitrelle® (Long Agonist Protocol) (N=13) | Gonal-f® + Ovitrelle® (Multi-dose Antagonist Protocol) (N=11)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Gene expression of the endometrium could not be analyzed due to poor quality of biopsy samples (poor mRNA quality) and poor recruitment in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other